CLINICAL TRIAL: NCT04199390
Title: Randomized Controlled Trial of Home-based Physical Therapy Versus Outpatient Clinic-based Physical Therapy Following Primary Anterior Total Hip Arthroplasty
Brief Title: Physical Therapy Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic One (Other)
Collaborators: Medacta USA (Industry)
Responsible Party: Principal Investigator, Thomas J Ellis, Principal Investigator, Orthopedic One
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20181607
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hip Osteoarthritis; Surgery
Keywords: total hip arthroplasty; physical therapy
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-based Physical Therapy (Active Comparator)
  Interventions: Procedure: total hip arthroplasty
- Home-based Physical Therapy (Active Comparator)
  Interventions: Procedure: total hip arthroplasty

INTERVENTIONS:
Procedure: total hip arthroplasty — each patient is expected to undergo an anterior total hip arthroplasty procedure and some sort of physical therapy postoperatively
  Other Names: physical therapy

SUMMARY:
130 patients undergoing primary unilateral total hip arthroplasty through anterior approach were enrolled and randomized into one of two groups. One group received standard of care clinic-based physical therapy postoperatively (clinic PT) while the other group underwent progressive home-based exercises to do after surgery (home PT). Patient surveys with Hip Osteoarthritis Outcome Scores (HOOS) and SF12v2 scores for both groups were obtained before surgery as well as 6, 14, and 24 weeks postop. Patients had the option to crossover into the other study group at their 6-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo primary unilateral anterior total hip arthroplasty for the treatment of arthritis under the care of the Principal investigator
* available for follow ups postoperatively

Exclusion Criteria:

* Age <18 or > 75
* Preoperative BMI ≥ 40
* Revision (i.e., non-primary) THA procedures
* Patients who have undergone THA in contralateral hip within the past 6 months
* Patient is scheduled for or anticipating THA on contralateral limb within 6 months
* Patients with an active infection (at the time of screening through surgery, as this is a surgical contraindication)
* Current co-morbidities such as alcohol or drug addiction, and/or mental disorders could potentially interfere with study participation
* Cognitive deficit or significant mental impairment that would, in the opinion of the investigator, impede patient self-reporting
* History of severe osteoporosis, metabolic bone disease, radioactive bone disease, or tumor in the bone surrounding the hip joint
* History of significant neurological and/or musculoskeletal disorders that may adversely affect gait after THA
* History of inflammatory hip arthritis
* History of septic hip arthritis in affected hip
* Patients requiring discharge to a rehabilitation center, skilled nursing facility, long-term care center, or convalescent home
* Non-English speaking
* Unable to give informed consent
* Currently enrolled in another therapeutic study for THA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Hip Disability and Osteoarthritis Outcome Scores | preoperative, postoperative 6 weeks, postoperative 12 weeks, and postoperative 24 weeks
Change in SF-12v2 Scores | preoperative and postoperative 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic One, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolford ML, Palso K, Bercovitz A. Hospitalization for total hip replacement among inpatients aged 45 and over: United States, 2000-2010. NCHS Data Brief. 2015 Feb;(186):1-8. PMID 25714040
- [Background] Ong KL, Lotke PA, Lau E, Manley MT, Kurtz SM. Prevalence and Costs of Rehabilitation and Physical Therapy After Primary TJA. J Arthroplasty. 2015 Jul;30(7):1121-6. doi: 10.1016/j.arth.2015.02.030. Epub 2015 Feb 28. PMID 25765130
- [Background] Kramer JF, Speechley M, Bourne R, Rorabeck C, Vaz M. Comparison of clinic- and home-based rehabilitation programs after total knee arthroplasty. Clin Orthop Relat Res. 2003 May;(410):225-34. doi: 10.1097/01.blo.0000063600.67412.11. PMID 12771834
- [Background] Galea MP, Levinger P, Lythgo N, Cimoli C, Weller R, Tully E, McMeeken J, Westh R. A targeted home- and center-based exercise program for people after total hip replacement: a randomized clinical trial. Arch Phys Med Rehabil. 2008 Aug;89(8):1442-7. doi: 10.1016/j.apmr.2007.11.058. Epub 2008 Jun 30. PMID 18586222
- [Background] Di Monaco M, Vallero F, Tappero R, Cavanna A. Rehabilitation after total hip arthroplasty: a systematic review of controlled trials on physical exercise programs. Eur J Phys Rehabil Med. 2009 Sep;45(3):303-17. Epub 2009 Feb 23. PMID 19238130
- [Background] Berger RA, Jacobs JJ, Meneghini RM, Della Valle C, Paprosky W, Rosenberg AG. Rapid rehabilitation and recovery with minimally invasive total hip arthroplasty. Clin Orthop Relat Res. 2004 Dec;(429):239-47. doi: 10.1097/01.blo.0000150127.80647.80. PMID 15577494
- [Background] Sharma V, Morgan PM, Cheng EY. Factors influencing early rehabilitation after THA: a systematic review. Clin Orthop Relat Res. 2009 Jun;467(6):1400-11. doi: 10.1007/s11999-009-0750-9. Epub 2009 Mar 10. PMID 19277807
- [Background] Austin MS, Urbani BT, Fleischman AN, Fernando ND, Purtill JJ, Hozack WJ, Parvizi J, Rothman RH. Formal Physical Therapy After Total Hip Arthroplasty Is Not Required: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Apr 19;99(8):648-655. doi: 10.2106/JBJS.16.00674. PMID 28419032